CLINICAL TRIAL: NCT02787070
Title: A Randomized Controlled Trial on Malaria Primaquine Treatment in Timika, Indonesia (TRIPI)
Acronym: TRIPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Timika Research Facility Kompleks RSMM, Timika-Papua, Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIPI
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Uncomplicated Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primaquine supervised (Active Comparator): 14 days of supervised primaquine treatment (0.5mg/kg/day).
  Interventions: Drug: PQ supervised
- Primaquine unsupervised (Active Comparator): 14 days of unsupervised primaquine treatment (0.5mg/kg/day).
  Interventions: Drug: PQ unsupervised

INTERVENTIONS:
Drug: PQ supervised
  Arms: Primaquine supervised
Drug: PQ unsupervised
  Arms: Primaquine unsupervised

SUMMARY:
Plasmodium vivax can form dormant liver stages that reactivate weeks or months following an acute infection. Recurrent infections can be associated with a febrile illness, a cumulative risk of severe anaemia, and even mortality. In co-endemic areas the risk of recurrence after both P. vivax and P. falciparum infections can be over 50% within 3 months. The only drug we have to kill P. vivax hypnozoites is primaquine which is currently given as a 14 day regimen. In Papua a retrospective study found very low effectiveness for unsupervised treatment. If true this has profound effects on treatment policy, suggesting that greater efforts are needed to encourage adherence to treatment.

We propose a cluster randomized, controlled, open label trial to assess the effectiveness of unsupervised versus supervised primaquine treatment in patients with uncomplicated malaria. Since the risk of recurrent P. vivax is high in patients with either P. vivax or P. falciparum, both infections will be included in the study. The study will be conducted in Mimika, in the southern part of Papua Province, Indonesia. Participants will be enrolled at village health posts and provided with schizontocidal treatment plus primaquine radical cure which will be either supervised or unsupervised depending on which cluster the clinic is in. Participants will be followed up for 6 months and assessed in regular intervals for the presence of patent and sub-patent malaria. The outcome of the study will contribute to an improved treatment scheme for uncomplicated malaria in this area.

ELIGIBILITY:
Inclusion Criteria:

* Infection with Plasmodium falciparum or P. vivax either alone or mixed
* Age >12 months
* Weight >5kg
* Living in the study clusters

Exclusion Criteria:

* General danger signs or symptoms of severe malaria
* Anaemia, defined as Hb <9g/dl
* G6PD deficiency (as determined by FST)
* Pregnant women as determined by Urine β-HCG pregnancy test
* Known hypersensitivity to any of the drugs given

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The incidence risk of symptomatic P. vivax malaria over 6 months in patients enrolled with any malaria infection | 6 months

SECONDARY OUTCOMES:
The incidence risk of symptomatic P. vivax malaria over 6 months in patients enrolled with P. vivax malaria infection | 6 months
The incidence risk of symptomatic P. vivax malaria over 6 months in patients enrolled with P. falciparum malaria infection | 6 months
The incidence rate of symptomatic P. vivax malaria over 6 months in patients enrolled with malaria due to P. falciparum or P. vivax | 6 months
The incidence rate of symptomatic P. vivax malaria over 6 months in patients enrolled with P. vivax malaria | 6 months
The incidence rate of symptomatic P. vivax malaria over 6 months in patients enrolled with P. falciparum malaria | 6 months
The incidence risk of patent or sub-microscopic P. vivax malaria over six months in patients enrolled with a malaria (sub-group analysis for patients recruited with P. vivax infection and P. falciparum infection) | 6 months
The incidence risk of any patent or sub-microscopic parasitaemia due to P. vivax or P. falciparum over six months in patients | 6 months
The proportion of patients vomiting their medication within 1 hour of administration | 1 hour
• The proportion of patients vomiting any of their primaquine doses during the 14 day supervised course | 14 days
• The proportion of adverse events and serious adverse events over 6 months in all patients | 6 months
• The incidence risk of severe anaemia (Hb<7g/dl) and/or the risk for blood transfusion over 6 months | 6 months
• The incidence risk of an acute drop in Hb >5g/dl within 14 days of starting primaquine treatment | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Timika Research Facility, Timika, Timika-Papua, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Poespoprodjo JR, Burdam FH, Candrawati F, Ley B, Meagher N, Kenangalem E, Indrawanti R, Trianty L, Thriemer K, Price DJ, Simpson JA, Price RN. Supervised versus unsupervised primaquine radical cure for the treatment of falciparum and vivax malaria in Papua, Indonesia: a cluster-randomised, controlled, open-label superiority trial. Lancet Infect Dis. 2022 Mar;22(3):367-376. doi: 10.1016/S1473-3099(21)00358-3. Epub 2021 Oct 25. PMID 34710363